CLINICAL TRIAL: NCT00004834
Title: Randomized Study of Cognitive-Behavioral Therapy vs Imipramine and Their Combination for Panic Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Long Island Jewish Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 199/13462; R10MH045963 (NIH); R10MH045965 (NIH); R10MH045964 (NIH); R10MH045966 (NIH)
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2013-02

CONDITIONS: Panic Disorder
Keywords: anxiety disorder; disease-related problem/condition; neurologic and psychiatric disorders; panic disorder; rare disease
MeSH Terms: conditions — Panic Disorder; Anxiety Disorders; Neurologic Manifestations; Mental Disorders; Rare Diseases | interventions — Imipramine; Cognitive Behavioral Therapy

INTERVENTIONS:
Drug: imipramine
Behavioral: cognitive-behavioral therapy

SUMMARY:
OBJECTIVES:

I. Determine which treatment is most effective for patients with panic disorder: cognitive-behavioral therapy (CBT) plus imipramine (IMI), CBT plus placebo, CBT alone, IMI alone, or placebo alone.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double-blind, placebo-controlled study. Patients are randomized to receive one of five treatments: cognitive-behavioral therapy (CBT) alone, imipramine plus medical management (IMI), CBT plus IMI, pill placebo plus medical management (PLA), or CBT plus PLA.

Patients are seen by therapists for 11 sessions over 12 weeks (3 sessions during days 1-10 followed by 6 weekly sessions and 2 biweekly sessions). Each CBT session lasts approximately 1 hour, each IMI session lasts approximately 30 minutes, and patients in combined treatment see 2 therapists for a total of about 80 minutes. Oral IMI or placebo is taken daily.

Patients not responding to placebo or IMI after the initial 12 weeks are offered alternative treatment for up to 3 months or given a referral; responders continue to be treated monthly for the next 6 months. This is followed by a washout period of 6 months, after which patients receive final assessment. All therapy and assessment sessions are video- or audiotaped.

Patients are interviewed by an independent evaluator at the start of treatment and 3, 9, and 15 months later, and must keep a set of weekly self-monitoring forms. In addition, patients complete rating forms and questionnaires, and undergo carbon dioxide measurement at the start of treatment and 3, 9, and 15 months later.

At study conclusion, patients are told which medication they received and receive treatment recommendations.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Principal diagnosis of panic disorder with or without mild agoraphobia, confirmed using the Anxiety Disorders Interview Schedule-Revised
* At least one full or limited panic attack per week within 2 weeks prior to initial assessment and 2 weeks prior to treatment

--Prior/Concurrent Therapy--

* Drug washout required if on anxiolytic or antidepressant medication No more than 10 benzodiazepine doses (0.5 mg alprazolam equivalent) within 2 weeks prior to treatment No more than 20 doses of benzodiazepine during baseline and acute treatment combined No more than one dose of benzodiazepine per day permitted
* No concurrent competing treatment

--Patient Characteristics--

* Not pregnant Negative serum pregnancy test required Effective contraception required of fertile women No psychotic, bipolar, or significant medical illnesses Not suicidal No significant substance abuse No prior nonresponse to either study treatment or related treatments No concurrent disability claims

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 326
Dates: Start 1998-05; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jack M. Gorman, Study Chair — Long Island Jewish Medical Center